CLINICAL TRIAL: NCT01867372
Title: Early Markers of Alzheimer's Disease in BLSA Participants: Structural and Functional Brain Changes
Brief Title: Early Markers of Alzheimer's Disease: Structural and Functional Brain Changes
Status: Terminated | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903328; 03-AG-N328
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2014-09-22

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

- Participants in the Baltimore Longitudinal Study of Aging are being studied to examine changes in brain structure and function over time, and to determine if these changes can predict the likelihood that an individual will develop thinking and memory impairments such as Alzheimer s disease later in life. Imaging studies and neuropsychological testing have been conducted on current participants, and new participants are being recruited to the study. To develop better treatments and therapies for aging-related memory loss and other disorders, researchers are interested in determining whether early prediction of thinking and memory impairments are accurate and in evaluating factors that affect these predictions.

Objectives:

- To use imaging studies and tests of thinking and memory to determine early markers of Alzheimer s disease and other cognitive impairments.

Eligibility:

- Current participants and new recruits to the Baltimore Longitudinal Study of Aging.

Design:

* Participants will be screened with a full medical history and physical examination, as well as blood and urine tests.
* Participants will have testing visits as directed by the study researchers. All participants will have tests as part of their an initial enrollment in the study, and may be asked to return yearly, 2 years later, or 4 years later for repeated tests.
* At each visit, participants will have brain imaging scans (including magnetic resonance imaging and/or magnetic resonance spectroscopy to measure brain structure and function, and positron emission tomography to study blood flow in the brain) to evaluate brain structure and function. Participants will also take tests of memory and problem-solving skills.
* Treatment will not be provided as part of this protocol.

DETAILED DESCRIPTION:
We are examining changes in brain structure and function as predictors of cognitive decline and impairment through longitudinal neuroimaging assessments of selected Baltimore Longitudinal Study of Aging (BLSA) participants. The hypothesis driving this study is that accelerated preclinical changes in brain structure and function in specific regions, including mesial temporal cortex, cingulate cortex, and inferior parietal cortex, will predict which individuals subsequently develop cognitive impairment and Alzheimer s disease. Since 1994, magnetic resonance imaging (MRI), positron emission tomography (PET), and neuropsychological testing have been performed for the neuroimaging participants, aged 55 and older. In the next phase of this study, we will continue longitudinal testing of older participants and will continue enrolling additional participants. We will continue MRI studies of brain structure, with enhanced measures of vascular changes, and will perform PET studies of cerebral blood flow, amyloid distribution in brain, and, in a subset of participants, cerebral glucose metabolism. We will also extend the MRI and neuropsychological evaluations to an additional 60 BLSA participants aged 20 to 54. Our initial data indicate substantial changes in brain volumes and tissue composition through the 5th evaluation, despite only minimal cognitive change in this generally healthy sample. We will continue to follow these individuals and will examine modifiers of both structural and functional brain changes and their associations with cognitive decline. Potential modulators include genetic factors, hormonal status and therapies, medications, dietary supplements, and other health-related factors. We have already observed acceleration of hippocampal volume loss in individuals at increased genetic risk for Alzheimer s disease, carriers of the apolipoprotein E epsilon 4 allele, and modulation of memory and regional cerebral blood flow activation patterns as a function of postmenopausal hormone therapy in women and endogenous testosterone concentrations in men. We will continue to examine these and other modifiers of brain-behavior associations. Early prediction of cognitive impairment and factors that alter the incidence or progression of disease will be essential as new therapies are on the horizon.

ELIGIBILITY:
* INCLUSION CRITERIA:

BLSA participants who do not meet exclusion criteria

EXCLUSION CRITERIA:

1. Miscellaneous: Body weight > 300 pounds, history of significant radiation exposure.
2. Participants with pacemakers, implanted electronic hearing devices, aneurysm clips, shrapnel, unallowed prosthetic or any other metallic device in their bodies.
3. Pre-existing CNS disease or severe cardiovascular disease (MI, CABG, angioplasty).

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2003-03-10; Primary Completion 2014-09-22 (Actual); Study Completion 2014-09-22

PRIMARY OUTCOMES:
Accelerated preclinical changes in brain structure and function in specific regions will predict which individuals develop cognitive impairment and Alzheimer s disease | Ongoing
Changes in brain structure are predictors of cognitive decline and impairment though neuroimaging assessments | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Resnick, Ph.D., Principal Investigator — National Institute on Aging (NIA)
Locations (3):
- United States (3):
  - Johns Hopkins University, Baltimore, Maryland
  - Kennedy Krieger Institute, Baltimore, Maryland
  - National Institute of Aging, Clinical Research Unit, Baltimore, Maryland